CLINICAL TRIAL: NCT01701219
Title: A Multicenter, 2-Cohort Study to Describe the Safety and Efficacy of Ceftaroline Fosamil in Subjects With Staphylococcus Aureus Bacteremia or With Persistent Methicillin-Resistant Staphylococcus Aureus Bacteremia
Brief Title: Safety and Efficacy Study of Ceftaroline in Subjects With Staphylococcus Aureus Bacteremia or With Persistent Methicillin-Resistant Staphylococcus Aureus Bacteremia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPT-MD-32
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Staphylococcus Aureus Bacteremia; Methicillin-resistant Staphylococcus Aureus (MRSA) Bacteremia
Keywords: Staphylococcus aureus bacteremia; Methicillin-resistant Staphylococcus aureus bacteremia; MRSA bacteremia; Blood; Adult; Infections; Blood Culture
MeSH Terms: conditions — Bacteremia; Infections | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Other): S. aureus on at least 1 blood culture within 72 hours of beginning study drug
  Interventions: Drug: Ceftaroline fosamil
- Cohort B (Other): MRSA on a baseline blood culture and on at least 1 additional blood culture after at least 72 hours of vancomycin and/or daptomycin treatment
  Interventions: Drug: Ceftaroline fosamil

INTERVENTIONS:
Drug: Ceftaroline fosamil — Ceftaroline fosamil 600 mg intravenous (IV) infused over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour) (dosing may be adjusted for renal function)
  Other Names: Teflaro®; PPI-0903; TAK-599; TAK599; PPI0903; Zinforo

SUMMARY:
This is a study of safety and efficacy of ceftaroline fosamil in Subjects with Staphylococcus aureus Bacteremia or with Methicillin-Resistant Staphylococcus aureus (MRSA) Bacteremia persisting after at least 72 hours of vancomycin and/or daptomycin treatment.

DETAILED DESCRIPTION:
Subjects with either S. aureus bacteremia or persistent MRSA bacteremia will be treated with open label ceftaroline fosamil, safety will be monitored and clearance of bacteremia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of bacteremia due solely to:

   * S. aureus on at least 1 blood culture within 72 hours of beginning study drug (Cohort A) OR
   * MRSA on a baseline blood culture and on at least 1 additional blood culture after at least 72 hours of vancomycin and/or daptomycin treatment (Cohort B).
2. Male or female ≥ 18 years of age.
3. If female of childbearing potential must be willing to practice sexual abstinence or dual methods of contraception during treatment and for at least 30 days after the last dose of study drug.
4. Expectation of survival for at least 2 months.

Exclusion Criteria:

1. For subjects in Cohort A: previous therapy for more than 48 hours with any parenteral antibiotic with activity against S. aureus within 72 hours of positive blood culture results.
2. For subjects in Cohort B: previous therapy for more than 48 hours with any parenteral antibiotic with activity against MRSA, except vancomycin and/or daptomycin, within 72 hours of positive blood culture results confirming persistence.
3. Previous episode of S. aureus bacteremia within 3 months.
4. Known left-sided endocarditis or prosthetic heart valve.
5. Osteomyelitis or prosthetic joint infection except new onset nonhardware-associated vertebral osteomyelitis.
6. History of any hypersensitivity or allergic reaction to any β-lactam antibacterial agent.
7. Evidence of significant hepatic, hematologic, or immunologic impairment.
8. Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of ceftaroline fosamil in adult Subjects (≥ 18 years of age) with Staphylococcus aureus Bacteremia or with MRSA Bacteremia persisting after at least 72 hours of vancomycin and/or daptomycin treatment | 60 days following completion of antibacterial therapy and discharge from the hospital, anticipated between 74 to 119 days
  Efficacy outcome measures:
  * Time to clearance of bacteremia
  * Time to defervescence
  * Clinical outcome
  * Mortality
  * Readmission

SECONDARY OUTCOMES:
Evaluate the efficacy of ceftaroline fosamil in adult Subjects (≥ 18 years of age) with Staphylococcus aureus Bacteremia or with MRSA Bacteremia persisting after at least 72 hours of vancomycin and/or daptomycin treatment | Between 3 and 119 days
  Safety evaluations will be conducted and assessments will include:
  * Adverse events including deaths will be evaluated
  * Laboratory: complete blood count (CBC) with differential and chemistry panel

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Sacramento, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Sylmar, California
  - Investigational Site, Torrance, California
  - Investigational Site, Hartford, Connecticut
  - Investigational Site, Pensacola, Florida
  - Investigational Site, Stuart, Florida
  - Investigational Site, Decatur, Georgia
  - Investigational Site, Macon, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Fort Wayne, Indiana
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Grosse Pointe Woods, Michigan
  - Investigational Site, Royal Oak, Michigan
  - Investigational Site, Laconia, New Hampshire
  - Investigational Site, Neptune City, New Jersey
  - Investigational Site, Newark, New Jersey
  - Investigational Site, Jamaica, New York
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Greenville, South Carolina
  - Investigational Site, Houston, Texas
  - Investigational Site, Annandale, Virginia
  - Investigational Site, Roanoke, Virginia

REFERENCES:
- See also: Sponsor Website — http://www.cerexa.com